CLINICAL TRIAL: NCT00003626
Title: Phase II Evaluation of Dolastatin-10 in Patients With Hormone Refractory Prostate Cancer
Brief Title: Dolastatin 10 in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Previous Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066708; P30CA022453 (NIH); WSU-D-1644; NCI-T98-0019
Record Dates: First submitted 1999-11-01; First posted 2004-08-17 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — dolastatin 10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dolastatin 10

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of dolastatin 10 in treating patients with metastatic prostate cancer that has not responded to previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate in patients with hormone refractory prostate cancer treated with dolastatin 10. II. Determine the toxicity of this regimen in this patient population.

OUTLINE: Patients receive dolastatin 10 IV bolus every 3 weeks. Treatment continues for a minimum of 2 courses in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Hormone refractory metastatic prostate cancer (stage D1 or D2) with no greater than 3 prior endocrine manipulations PSA level increased on 3 consecutive measurements at least 2 weeks apart PSA at least 10 ng/mL (not required if measurable disease)

PATIENT CHARACTERISTICS: Age: Not specified Performance status: SWOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count at least 1,500/mm3 Hemoglobin at least 8 g/dL Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2 mg/dL AST no greater than 2 times upper limit of normal Renal: Creatinine less than 2.0 mg/dL Other: No other serious medical illness No serious infection No other prior malignancy within the past 5 years except nonmelanoma skin cancer or any in situ carcinoma

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: See Disease Characteristics Concurrent LHRH-agonist therapy allowed without antiandrogens At least 4 weeks since prior flutamide and nilutamide At least 6 weeks since prior bicalutamide At least 4 weeks since other prior hormone therapy including steroids Radiotherapy: At least 4 weeks since prior radiation therapy and recovered No prior strontium Surgery: Recovered from prior surgery

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-10; Primary Completion 1999-12 (Actual); Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hadi A. Hussain, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Denver, Colorado
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Vaishampayan U, Glode M, Du W, Kraft A, Hudes G, Wright J, Hussain M. Phase II study of dolastatin-10 in patients with hormone-refractory metastatic prostate adenocarcinoma. Clin Cancer Res. 2000 Nov;6(11):4205-8. PMID 11106233